CLINICAL TRIAL: NCT00299637
Title: Changes in Blood Flow in MCA of Fetuses to Mothers Having Clinical Chorioamnionitis During Labor Comparing to Fetuses to Healthy Mothers.
Brief Title: Changes in Blood Flow in MCA of Fetuses to Mothers Having Clinical Chorioamnionitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: MCA chorioamnionitis HMO-CTIL
Record Dates: First submitted 2006-03-05; First posted 2006-03-07 (Estimated); Last update posted 2006-11-30 (Estimated); Status verified 2006-03

CONDITIONS: Chorioamnionitis
MeSH Terms: conditions — Chorioamnionitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
This study will try to determine whether fetuses to mothers having clinical chorioamnionitis have changes in blood flow in middle cerebral artery.

DETAILED DESCRIPTION:
This study will try to determine whether fetuses to mothers having clinical chorioamnionitis have changes in blood flow in middle cerebral artery.

MCA flow parameters will be evaluated during labor of women with and wthout chorioamnionitis

ELIGIBILITY:
Inclusion Criteria:

* women giving birth week 37-42
* healthy
* one fetus

Exclusion Criteria:

* more than one fetus
* IUGR
* illness or damage to fetus

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2006-10; Study Completion 2007-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: David Mankuta, MD, Study Chair — Hadassah Medical Organization
Locations (1):
- Haddasah Medical Organization, Jerusalem, Israel